CLINICAL TRIAL: NCT01549548
Title: Treatment Plan for the Compassionate Use of Ponatinib (AP24534) in Patients With Imatinib-, Dasatinib-, and Nilotinib- Resistant/Intolerant Philadelphia Chromosome Positive Leukemias.
Brief Title: Compassionate Use Ponatinib
Status: No longer available | Type: Expanded Access
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00008238
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Philadelphia Chromosome Positive (Ph+) Leukemias; Chronic Myeloid Leukemia
Keywords: CML
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

INTERVENTIONS:
Drug: Ponatinib — Patients will receive Ponatinib 45 mg by mouth as a single daily dose on an empty stomach (no food 2 hours prior to and after dosing) on day 1 and continuous once-daily dosing everyday thereafter. Each patient will receive daily Ponatinib until disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: AP24534

SUMMARY:
The main purpose of this protocol is to provide expanded access to the study drug (Ponatinib/AP24534) for people with imatinib-, dasatinib-, and nilotinib- resistant/intolerant Philadelphia Chromosome Positive (Ph+) Leukemias. The other purpose of this protocol is to monitor the safety of the study drug in people with Ph+ Leukemias that have not responded to prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Cytogenetic or PCR-based diagnosis of any phase of Ph+ acute lymphoblastic leukemia (ALL) and documented resistance or intolerance to imatinib and a second TKI (nilotinib, dasatinib, bosutinib)
* Eastern Cooperative Oncology Group(ECOG) performance status of 0-2
* Washout from prior anti-proliferative or anti-leukemia treatment: 3 days for hydroxyurea/anagrelide and tyrosine kinase inhibitors
* < Grade 2 or baseline recovery from prior therapy related toxicities (except alopecia)
* At least 3 months post allogeneic stem cell transplantation
* Able to take oral capsules reliably
* AST/ALT less than or equal to 2.5 times ULN, or less than 5 times ULN if attributable to involvement of leukemia
* No active clinical or radiographic pancreatitis
* At least 18 years of age
* Willingness of male and female subjects to use reliable methods of birth control (when applicable)

Exclusion Criteria:

* Subjects with Philadelphia Chromosome and BCR-ABL-negative chronic myeloid leukemia (CML)
* Major surgery or radiotherapy within 7 days before the first dose of Ponatinib (recovery from any previous surgery should be complete before day 1)
* Clinically significant active/uncompensated or uncontrolled cardiac disease (active congestive heart failure; uncontrolled angina or hypertension; myocardial infarction in the past 3 months; clinically significant untreated ventricular arrhythmia; diagnosed or suspected congenital or acquired prolonged QT syndrome; unexplained syncope; history of prolonged QTc)
* Prolonged QTc (> 0.48 sec)
* Pregnant or breastfeeding women
* Evidence of serious active infection, or significant medical or psychiatric illness
* Known seropositivity to HIV, or current acute or chronic Hepatitis B or Hepatitis C (antigen positive), cirrhosis, or clinically significant abnormal lab finding that would, in the investigator's judgment, make the subject inappropriate for this study
* Prior resistance to Ponatinib

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States